CLINICAL TRIAL: NCT05532748
Title: Distribution of Pulmonary Ventilation With the Modified Pachon Incentive vs. Another Branded Respiratory Incentive, Through Electrical Impedance Tomography, in a Healthy Volunteers of the City of Cali
Brief Title: Distribution of Pulmonary Ventilation With the Modified Pachon Incentive vs. Branded Respiratory Incentive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad del Valle, Colombia (Other)
Responsible Party: Principal Investigator, Esther Cecilia Wilches Luna, Full professor, Universidad del Valle, Colombia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 031-022
Record Dates: First submitted 2022-08-29; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Ventilation
Keywords: Tomography; Electric Impedance; Spirometry; Respiratory Therapy; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: The objective of this research is to compare the distribution of pulmonary ventilation using Electrical Impedance Tomography during the use of the Incentivo Modificado de Pachón and a commercial respiratory incentive, in healthy adults from the City of Cali (Colombia), for which A sample of 20 healthy subjects (10 men and 10 women) between 18 and 65 years of age will be used, who, after meeting the selection criteria, will undergo the first ventilation measurement using EIT with the incentive that has been randomly assigned to the participant, The second measurement will be carried out one week after the first measurement with the other incentive has been carried out, to complete the washout period, both measurements will be carried out by the principal investigator.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor of results will be masked, the data will be delivered encrypted with a code for the analysis of the measurement of each of the respiratory incentives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Pachon's incentive, then Branded incentive "Triflo II®" (Experimental): The first measurement with the tomograph will be made using the modified Pachon's incentive, and a week later the measurement will be made using the branded incentive
  Interventions: Device: Respiratory exercise protocol with the modified Pachon's incentive; Device: Respiratory exercise protocol with Branded respiratory incentive, "Triflo II®"
- Branded incentive "Triflo II®", then modified Pachon's incentive (Active Comparator): The first measurement with the tomograph will be made using the branded incentive, and a week later the measurement will be made using the modified Pachon's incentive.
  Interventions: Device: Respiratory exercise protocol with the modified Pachon's incentive; Device: Respiratory exercise protocol with Branded respiratory incentive, "Triflo II®"

INTERVENTIONS:
Device: Respiratory exercise protocol with the modified Pachon's incentive — With the participant sitting on a chair, with their back against the backrest, they will hold the device with the hand that is most comfortable for them and place the mouthpiece in their mouth, ensuring a correct seal with their lips.
  You will be asked to take a slow, deep breath, fully stretching the condom, and hold your breath for at least 5 seconds. Expiration will be performed passively through the device without removing it from the mouth and without performing any forced maneuver.
  There will be 3 series of 10 breaths with a 1-minute rest between series. The total number of breaths for the entire session will be 30; the maneuver will end once the series and repetitions are finished. You will be asked to remove the mouthpiece from your mouth and breathe for 3 minutes at a gentle intensity through your nose without extra effort.
  All these instructions will be explained through a video.
  Other Names: IMP
Device: Respiratory exercise protocol with Branded respiratory incentive, "Triflo II®" — With the participant sitting on a chair, with their back against the backrest, they will hold the device with the hand that is most comfortable for them and place the mouthpiece in their mouth, ensuring a correct seal with their lips.
  You will be asked to take a smooth deep breath lifting as many spheres as you can and hold your breath for at least 5 seconds. Expiration will be performed passively through the device without removing it from the mouth and without performing any forced maneuver.
  There will be 3 series of 10 breaths with a 1-minute rest between series. The total number of breaths for the entire session will be 30; the maneuver will end once the series and repetitions are finished. You will be asked to remove the mouthpiece from your mouth and breathe gently through your nose for 3 minutes without extra effort.
  All these instructions will be explained through a video.
  Other Names: Triflo II®

SUMMARY:
Incentive spirometry is a method to stimulate deep breathing and maximum sustained inflations, which provides participants with visual feedback on the inspiratory volume achieved, favoring lung inflation. Its multiple benefits and ease of use favor adherence, making it a common device used in the clinical environment.

This device is used in pathologies or procedures that can cause decreased function and respiratory mechanics, such as thoracoabdominal surgeries, and is indicated to reduce the incidence of postoperative pulmonary complications. It is also indicated in the presence of pulmonary atelectasis or conditions that predispose to the development of pulmonary atelectasis, in patients with prolonged bed rest, patients with neuromuscular disease, patients with spinal cord injury, and patients undergoing coronary bypass, among others.

In 2004, students from the Universidad del Valle carried out an investigation whose result was the creation of the Incentivo Modificado de Pachon, a handcrafted design device that allows mobilizing flows ranging from 600 CC/sec to more than 1400 CC/sec, which characterizes it as a flow respiratory incentive.

In 2020, the device obtained the endorsement of the Superintendence of Industry and Commerce, however, to date no studies have been carried out that objectively verify the effect that the modified Pachon's incentive (Incentivo Modificado de Pachon by the name in Spanish) has on the distribution of ventilation in comparison with another Branded respiratory incentive.

Electrical Impedance Tomography is a diagnostic tool that, employing a belt of electrodes connected around the user's chest, uses the electrical characteristics of the tissue, to provide information in a non-invasive, continuous way, on foot. bedside and radiation-free on pulmonary ventilation and perfusion, as it allows repeated imaging of tidal volume distribution, as well as distinguishing the characteristic regional filling and emptying of each lung, all in real-time and safely.

In this study, the distribution of pulmonary ventilation between the modified Pachon's incentive vs. another Branded respiratory incentive will be compared, through electrical impedance tomography, in a healthy population of the city of Cali.

The hypothesis to be tested is that the distribution of Pulmonary ventilation measured by Electrical Impedance Tomography is similar between the modified Pachon's incentive and another Branded flow respiratory incentive.

DETAILED DESCRIPTION:
The variables to be measured are:

Main variables:

* EELI Delta (ΔEELI): Measures the change in the average end-expiratory pulmonary impedance before and after an intervention
* MTV ROI: Minute regional tidal variation

Secondary variables:

* IPAQ: Instrument that provides information on estimated energy expenditure in 24 hours in the different areas of daily life
* Charlson index: Relates long-term mortality with the participant's comorbidity
* %FEV1 pred: Percentage of the predicted forced expired volume in the first second
* %FVC pred: Percentage of predicted forced vital capacity
* %FVC/FEV1: Percentage of predicted of relationship between forced vital capacity and FEV1
* Labor Occupation: Includes the labor function of the worker
* Level of schooling: the highest level of studies completed or in progress
* Marital status: situation determined by your family relationships, from marriage or kinship
* Socioeconomic Stratum: Classification in strata of residential properties
* Personal history: Compilation of information on the health of the person and pathologies that he/she suffers from
* Height: Measurement of the height of the human body from the feet to the roof of the cranial vault
* Weight: Force with which bodies are attracted towards the center of the earth by the action of gravity
* BMI: Relationship between weight and height
* Heart rate: Number of times the heart contracts in one minute
* Respiratory rate: Number of breaths in one minute
* Oxygen Saturation: Measurement of the amount of oxygen available in the blood
* Dyspnea: Difficulty breathing

Materials and Instruments:

The instruments that will be used in the study will be: Height rod, scale, Spirometer, Incentivo Modificado de Pachon, Hudson Flow Respiratory Incentive, equipment to measure impedance (Pulmovista), and data collection format. These are described below:

* Modified Pachon's incentive (Incentivo Modificado de Pachon by the name in Spanish): handmade device that imitates conventional respiratory incentives, but is made with recyclable, low-cost materials and is also easy to manufacture. Modified in 2004 in a research project by students from the Universidad del Valle, they defined that the Modified Pachon's incentive allows for the mobilization of flows that oscillate between 600 cc/sec up to more than 1400 cc/sec which characterizes it as a flow incentive. The materials used for its construction are a non-lubricated buretrol and a Today brand condom
* Triflo® II Respiratory Incentive: A method of encouraging deep voluntary breathing, which provides participants with visual feedback on inspiratory volume, employing 3 color-coded balls in three chambers, with a mouthpiece and tube. The minimum flow is marked on each chamber: 600, 900, and 1200 ml/Seg.. It is manufactured by HUDSON RCI
* PulmoVista 500®: it is an electrical impedance tomograph, from Dräger. The data is continuously represented in the form of images, curves, and parameters to observe ventilation continuously and directly in various lung regions, as well as the changes that occur in lung volumes at the end of expiration, non-invasively, in time. real and directly next to the bed
* Spirometer: This is a device that is commonly used to assess how well the lungs are working by measuring how much air you breathe in, how much you breathe out, and how quickly you breathe out. Spirometry is used to diagnose asthma, chronic obstructive pulmonary disease, and other diseases that affect breathing. For this study, a medgraphics cardiorespiratory diagnostics® brand spirometer will be used, which works with the breeze suite 6.4.1.44 SP4 system
* Stadiometer: it is a height meter that is fixed to the wall or support and is used to accurately measure people, so that when it is placed under it, the stadiometer will rest on their head, indicating the height on the dial. exactly who is using it. For this study, a SECA model 213® stadiometer will be used
* Scale: Device used to measure weights. For this study, a SECA® brand scale will be used

For this research, a data collection format was designed:

• Format created by the researcher consisting of a section on sociodemographic information, personal and family history, anthropometric data, level of physical activity, lung function data and results on ventilation and global and regional lung impedance for each individual

To measure clinical stability and the level of physical activity, the following instruments will be used:

* Charlson index: it is a life expectancy evaluation system, depending on the age at which it is evaluated, and the subject's comorbidities. In addition to age, it consists of 19 pathology items with their respective rating, which, if present, have been found to have a specific influence on the subject's life expectancy
* International Physical Activity Questionnaire (IPAQ) short version: IPAQ researchers developed several versions of the instrument according to the number of questions (short or long). The short version consists of 7 items and provides information about the time the person spends performing moderate and vigorous intensity activities, walking and sitting The research will be carried out in four stages: Preparation for the study, design, and adjustment of instruments, data collection, and data analysis. Ordered according to the logical steps to follow within the development of obtaining the required data

Phase 1: Preparation for the study At this stage, the search for initial information will be carried out, for this a bibliographic review will be carried out for the present study that includes research published in different databases, related to the validation and comparison of medical devices, the use of electrical impedance tomography and studies related to the use of respiratory incentive in the clinical setting and their levels of evidence. Once this is done, the research approach, the study design, the form of selection and sample size, and the writing of the document will be carried out For the development of this study, the main researcher will carry out 24-hour training in the handling of the equipment with expert personnel in its handling The informed consent will be designed and the written research work will be sent to the ethics committee to receive the endorsement

Phase 2: Design and adjustment of instruments The data collection instrument will be designed For the standardization of anthropometric measurements (weight and height), Standardized Operating Procedures 1 and 2 will be used For the measurement of electrical impedance tomography, Standard Operating Procedures 3, designed for projects previously carried out by the GIESC research group, will be used. "Effect of two lung reexpansion techniques on the ventilation of participants undergoing cardiovascular surgery. Controlled clinical trial phase II b" The pilot test will be carried out with 5 healthy subjects who will not be part of the sample, they will be informed about the research, they will be asked to sign the informed consent and the measurements and data collection will be carried out with the designed data collection format. by the researcher

Phase 3: Data Collection:

* Call for participants For the recruitment of healthy volunteers between 18-65 years of age in the community of Santiago de Cali, direct contact will be made with people from the administrative areas of the Universidad del Valle, from the research groups of the Universidad del Valle, family and friends who will initially be provided with information about the objectives of the research and will be invited to participate The electrical impedance tomography will be performed in the movement laboratory located in the health faculty of the Universidad del Valle and the spirometries will be performed at the Hospital Universitario del Valle
* Data collection protocol:

  * Performance of spirometry This measurement will be carried out at the Hospital Universitario del Valle, it will be carried out by the researcher, who is a physiotherapist specializing in cardiopulmonary physiotherapy. The day of the test will begin with the completion of the informed consent, this will be read and explained to the participant and will continue to the signature. On this day, the researcher will fill out the sociodemographic data of the participant, weight and height measurement, Charlson index, and IPAQ abbreviated questionnaire, according to the instructions defined in the Standard Operating Procedures designed for each one, in the data collection format Spirometry will be performed according to the institutional protocol of the Hospital Universitario del Valle. The duration of this procedure will take approximately 1 hour
  * Randomization The randomization to choose which will be the first device that each participant will use and to which the first ventilation measurement will be carried out using electrical impedance tomography will be carried out by simple randomization The first measurement will be carried out with the incentive that has been randomly assigned to the participant, the second measurement will be carried out one week after the first measurement has been carried out with the other incentive, with the objective that the washing period is fulfilled, both measurements will be carried out by the principal investigator For the measurement of the Electrical Impedance Tomography, a standardized operating procedure will be carried out, and for the application of the protocol for the use of respiratory incentives, the instructions defined in the standardized operating procedures carried out for their use will be followed. The duration of this procedure will be approximately 30 minutes for each measurement
  * Moments of electrical impedance tomography measurement

Once the patient is connected to the tomograph, once it is verified that it is being measured properly, that the patient is well positioned and that the signal is of high quality, the recording will begin. tomograph record; After the first two minutes of calm breathing have elapsed, the first event will be marked, which will be recorded as "pre", and the use of the corresponding respiratory incentive will begin. The proper use of the device will be previously explained to you through a video that will illustrate the correct way to use it. The participant will receive visual feedback from the device when the condom is raised within the buretrol in the case of the Modified Pachon's incentive or when the spheres are raised in the branded incentive Three series of ten breaths will be performed, with a 1-minute rest between series. In the last repetition of the third series, the second event will be marked, which will be recorded as "intra" The maneuver will be finished once the series and repetitions are finished, removing the mouthpiece from the participant's mouth and they will be asked to continue breathing calmly for 2 minutes, after which the third event will be marked, which will be recorded as "post". And the recording of the record will be terminated At the beginning and the end of the intervention, clinical data will be taken (heart rate and oxygen saturation) and 2 minutes after finishing the test The session may be interrupted if the participant does not wish to continue with the intervention, if the participant shows intolerance to the maneuver After each measurement is finished with each participant, the equipment will be disinfected

o Quality Control

1. To guarantee the quality of the registered information, the main investigator will carry out random reviews in which he will corroborate the coherence between the original information of the tomographer, that of the registration in the formats and that of the database. The detected errors will be corrected
2. An external person to the study, who will not participate in the measurements, will randomly review the formats once every 15 days to verify the information before entering it into the database. Additionally, once a month a meeting will be held with the research group to socialize project progress

ELIGIBILITY:
Inclusion Criteria:

* People aged between 18-65 years
* People with clinical stability, defined as the absence of any acute illness during the previous 6 weeks and a Charlson index score of 0-1 (12% mortality/year- no comorbidity)
* People with body mass index (BMI) 18.5 - 35 Kg/m2
* People without mental or cognitive alterations
* People who accept informed consent

Exclusion Criteria:

* People with pacemakers, cardioverters or cardio defibrillators.
* People with metal implants
* People with any condition in which the registration in the CT scanner signal is low.
* Women in pregnancy
* Participants with injuries, skin changes or presence of devices that prevent the placement of the electrode belt around the chest.
* People with a high level of physical activity according to the IPAQ questionnaire short version
* People whose spirometry registers obstruction or restriction
* People who do not understand the verbal command of the incentive technique

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
EELI Delta (ΔEELI) | Event 1 "pre": after the first 2 minutes of calm breathing. Event 2 "intra": In the last repetition of the third series of the use of the device. Event 3 "post": 2 minutes after finishing the three series of 10 repetitions
  Measures the change in the average end-expiratory pulmonary impedance between before and after an intervention.
  Measurement Unit: Arbitrary Impedance Units (A.U)
MTV ROI | Event 1 "pre": after the first 2 minutes of calm breathing. Event 2 "intra": In the last repetition of the third series of the use of the device. Event 3 "post": 2 minutes after finishing the three series of 10 repetitions
  Minute regional tidal variation. Measurement Unit: Arbitrary Impedance Units (A.U)

SECONDARY OUTCOMES:
Heart rate | after two minutes of calm breathing, after two minutes of the use of each respiratory incentive
  It is the number of times the heart contracts in one minute.
Oxygen saturation | after two minutes of calm breathing, after two minutes of the use of each respiratory incentive
  A measure of the amount of oxygen available in the blood Measurement unit: percentage, from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Noraelena Mera Quintero, Pt, MsC(c), Principal Investigator — universidad del Valle; Esther C Wilches Luna, Pt, PhD, Study Director — Universidad del Valle; Vicente A Benavides Cordoba, Pt, PhD, Study Director — Universidad del Valle
Locations (1):
- Universidad del Valle, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Yes
all collected individual participant data
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: from January 2023 to January 2033
Access Criteria: for future publications or for the development of subsequent projects

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT05532748/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT05532748/ICF_001.pdf